CLINICAL TRIAL: NCT05938348
Title: Pain Relief Effect of Angiopuncture for Patients With Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111111
Record Dates: First submitted 2023-06-07; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pain scores of patients before and after (6h, 12h, 24h, 48h, 72h) angiopuncture. (Experimental): investigators done angiopuncture on perforators in human. Pain score will be assessed on both before and after the treatment.
  Interventions: Behavioral: angiopuncture

INTERVENTIONS:
Behavioral: angiopuncture — we conducted acupuncture on perforators by using acupuncture needles.

SUMMARY:
The study aimed to investigate the effectiveness of angiopuncture therapy in pain alleviation for postoperative pain patients. The study involved patients aged 20-65 with acute foot and ankle trauma and pain after surgery. Physicians used handheld ultrasound Doppler to measure perforators, puncture participants with a filiform needle, and monitor pain scores and heart rate data before and after acupuncture. The duration of therapy was 20 minutes per day for 72 hours, with pain measured using the numerical rating scale. The study aimed to compare the outcomes before and after angiopuncture.

DETAILED DESCRIPTION:
In order to give therapeutic therapy, solid filiform needles are inserted into the skin during dry needling (DN), traditional acupuncture (TA), and western medical acupuncture (WMA). DN is a treatment used to treat painful musculoskeletal illnesses, whereas TA and WMA have a wider variety of indications, including musculoskeletal discomfort, gastrointestinal problems, and neurological concerns. While DN implants are used in trigger points, acupuncture is for acupoints.

In addition, common methods include injections of painkillers, oral medications, and nerve blocks. Angiopuncture therapy is being used for the first time as a method of pain management in this article. The aim was to investigate if skin perforating needling therapy could alleviate postoperative pain in patients.

Patients with recent foot and ankle surgery who have had acute foot and ankle injuries and pain. Doctors measured three to four perforators at the proximal end of the trauma site using a handheld ultrasound Doppler, punctured the perforators for 15 minutes with a filiform needle (size: 0.18mm gauge * 25mm length), and then monitored the patient's pain level and heart rate data before and after acupuncture Variety. If pain relief is possible, they'll do it. Risks include becoming more painful.

To create numbers, investigators employed an internet table generator. Despite having just one group, investigators compared the results of angiopuncture before and after therapy lasts for 20 minutes per day for 72 hours. Numeric rating scale (NRS) pain score at baseline: 6, 12, 24, 36, 48, 60, and 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* aged 20-65 years
* acute foot or ankle trauma
* pain after foot or ankle surgery

Exclusion Criteria:

* Have scars and deformities on the lower extremity surface
* cannot cooperate with the locating method of angiopuncture
* allergy to any material
* pregnant women
* breastfeeding women

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Participants reporting a score based on Numeric Pain Rating Scale | 6 hours after surgery
  A score was reported by participants based on the Numeric Pain Rating Scale. The lowest score is 0, and the highest score is 10. Higher scores mean a worse outcome which is more painful.
Participants reporting a score based on Numeric Pain Rating Scale | 12 hours after surgery
  A score was reported by participants based on the Numeric Pain Rating Scale. The lowest score is 0, and the highest score is 10. Higher scores mean a worse outcome which is more painful.
Participants reporting a score based on Numeric Pain Rating Scale | 24 hours after surgery
  A score was reported by participants based on the Numeric Pain Rating Scale. The lowest score is 0, and the highest score is 10. Higher scores mean a worse outcome which is more painful.
Participants reporting a score based on Numeric Pain Rating Scale | 36 hours after surgery
  A score was reported by participants based on the Numeric Pain Rating Scale. The lowest score is 0, and the highest score is 10. Higher scores mean a worse outcome which is more painful.
Participants reporting a score based on Numeric Pain Rating Scale | 48 hours after surgery
  A score was reported by participants based on the Numeric Pain Rating Scale. The lowest score is 0, and the highest score is 10. Higher scores mean a worse outcome which is more painful.
Participants reporting a score based on Numeric Pain Rating Scale | 60 hours after surgery
  A score was reported by participants based on the Numeric Pain Rating Scale. The lowest score is 0, and the highest score is 10. Higher scores mean a worse outcome which is more painful.
Participants reporting a score based on Numeric Pain Rating Scale | 72 hours after surgery
  A score was reported by participants based on the Numeric Pain Rating Scale. The lowest score is 0, and the highest score is 10. Higher scores mean a worse outcome which is more painful.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaomi People'S Hospital, Gaomi, Shandong, China

REFERENCES:
- [Derived] Han R, Feng W, Guo C, Ding Z, Hu J. Pain relief effect of angiopuncture therapy on patients with postoperative pain: A clinical trial. Medicine (Baltimore). 2024 Jan 12;103(2):e36847. doi: 10.1097/MD.0000000000036847. PMID 38215127